CLINICAL TRIAL: NCT07122830
Title: From Intention to Implementation: Evaluating the Feasibility and Acceptability of Family Integrated Care in Special Care Nursery
Brief Title: Family Integrated Care: A Feasibility Study in a Level II Special Care Nursery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Chan Shu Hui, Principal Investigator, KK Women's and Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-2643; CRADLE/2023/RES/003 (Other Grant/Funding Number: Paediatric Academic Clinical Programme)
Record Dates: First submitted 2025-07-20; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Family Centered Care; Neonatal
Keywords: Feasibility; Family Integrated Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIC Group (Active Comparator)
  Interventions: Other: Family Education and Parental Involvement
- Control Group (No Intervention): The usual standard of care will be provided for this group.

INTERVENTIONS:
Other: Family Education and Parental Involvement — Parents will be oriented to the programme, tools provided for their own learning (pamphlets, information handouts, audio-visual resources), and a checklist of infant care topics to be completed. The primary caregiver will be asked to commit to spending one to two hours per day to attend education sessions on the topic(s) of their choice. Parents will be encouraged to provide progressively more daily care for their infants as they complete more education sessions. After each education session, parents will check off for each completed topic on their skills checklist.
  Arms: FIC Group

SUMMARY:
The goal of this mixed methods study is to assess the feasibility and acceptability of a parent-led family integrated care program in a Level II neonatal unit.

The main questions it aims to answer are:

* Is it feasible to implement a parent-led Family Integrated Care (FIC) program in a Level II neonatal unit?
* How acceptable is the FIC program to parents and nurses?
* Can the FIC program help improve parental self-efficacy and infant outcomes?

ELIGIBILITY:
Inclusion Criteria:

* Parents of infants admitted to the Level II neonatal unit who anticipate at least 2 weeks of stay
* Parents of infants who can commit to coming daily for one to two hours.

Exclusion Criteria:

* Infants have severe congenital anomalies
* Infants receiving pallitaive care
* Infants who are critically ill / deemed unlikely to survive
* Infants scheduled for early transfer
* Parents are unable to participate due to health, social, or language issues that would inhibit their communication with the medical and nursing team.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Through grant period, up to 6 months
  This study will examine the length of time taken to complete participant recruitment, and recruitment rates.
Retention Rates | Up to 6 months
  This will be evaluated by examining the participants drop-out rates throughout the study. This will be used to assess the fidelity of the program.
Completion of FIC program | Through grant period, up to 6 months
  This will be evaluated by examining the percentage completion of the FIC program teaching sessions by each participant. This will be used to assess the fidelity of the program.
Parent Experience of FIC Program | Through grant period, up to 6 months
  Parents will have a semi-structured interviews to have a qualitative evaluation of their experience of the FIC program. This study aims to identify any barriers and/or facilitating factors of the program.
Nurses' Experience of the FIC Program | Up to 1 year
  Nurses will have a quantitative and qualitative evaluation of the program through a post-implementation survey and focused group discussion respectively. This study aims to identify any barriers and/or facilitators through their experience.
  The nurses' survey consists of 8-items, scored on a 5-point Likert scale. Nurses can score between 8 - 40, with a higher score reflecting a better experience of the FIC program.

SECONDARY OUTCOMES:
Parental Self-Efficacy | Through grant period, up to 6 months
  Parents will complete the Perceived Maternal Parenting Self-Efficacy (PMPS-E) Questionnaire pre-test and post-test to evaluate for improvements in their self-efficacy after going through the intervention.
  The PMPS-E Questionnaire is a 20-item questionnaire that uses a 4-point Likert scale ranging from 'Strongly Disagree' (Score = 1), 'Disagree' (Score = 2), 'Agree' (Score = 3), and 'Strongly Agree' (Score = 4). Participants can score between 20 to 80, where a higher score reflects higher self-efficacy.
Frequency of Parental Visits | Through grant period, up to 6 months
  This study aims to evaluate whether parents in the FIC group have a higher frequency of visits, measured in number of days, compared to those in the control group.
Frequency of Kangaroo Care | Through grant period, up to 6 months
  This study aims to evaluate whether parents in the FIC group have practice kangaroo care more often, measured in number of times done, compared to those in the control group.
Duration of Kangaroo Care | Through grant period, up to 6 months
  This study aims to evaluate whether parents in the FIC group carry our kangaroo care for longer periods of time, measured in number of minutes, compared to those in the control group.
Frequency of Breastfeeding | Through grant period, up to 6 months
  This study aims to assess whether mothers in the FIC group engage in more breastfeeding, as measured by the number of feeds, compared to those in the control group.
Duration of Breastfeeding | Through grant period, up to 6 months
  This study aims to assess whether mothers in the FIC group engage in longer breastfeeding sessions, measured by the number of minutes, compared to those in the control group.
Length of Stay | Through grant period, up to 6 months]
  This study aims to evaluate whether infants in the FIC group have a shorter length of stay, measured in the number of days, compared to the control group.
Infants Weight Gain | Through grant period, up to 6 months
  This study aims to assess whether infants in the FIC Group have higher weight gain compared to infants in the control group. The infants' birth weight and weight at discharge, measured in grams, will be collected and calculated [discharge weight (g) - birth weight (g)] to derive the infants' weight gain (g).
Nasogastric Tube Retention Time | Through grant period, up to 6 months
  This study aims to assess whether infants in the FIC group are able to achieve full oral feeding earlier than infants in the control group. This will be evaluated using the duration of their nasogastric tube retention time, measured in the number of days.

CONTACTS AND LOCATIONS:
Overall Officials: Shu Hui Chan, BSc (Nursing) (Honours), Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: CSR
Time Frame: IPD and supporting information will be stored and available for 10 years from 24 April 2025 until 1 April 2035. Thereafter, the stored IPD will be deleted and destroyed in accordance with PDPA guidelines of the hospital.
Access Criteria: Only the principle investigator will be able to access it via an encrypted access to the excel spreadsheet.